CLINICAL TRIAL: NCT03847454
Title: A Personal Mobility Device for Elderly Physical Rehabilitation: a Study of Acceptance and Efficiency
Brief Title: REACH Personal Mobility Device Testing
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Prof. Antoine Geissbuhler, Chair of the division of eHealth and telemedicine, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-01516
Record Dates: First submitted 2019-01-29; First posted 2019-02-20 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Musculoskeletal Diseases or Conditions; Rehabilitation
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention REACH group (Experimental): The intervention REACH consists of a mobility device called ActivLife developed by Alreh Medical, that is coupled with serious games, a Kinect sensor and a wearable sensor called Stepwatch, to continuously measure the patients physical activity. The participants will receive 30 min training every day during 3 weeks. 3 times a week the standard training will be replaced with the intervention. The training is conducted/ supervised by a physiotherapist.
  Interventions: Combination Product: REACH
- Control group (Standard of care) (Active Comparator): The participants will receive the standard of care as intervention which consists of 30 min training every day during 3 weeks. The training is conducted by a physiotherapist.
  Interventions: Other: Standard of care

INTERVENTIONS:
Combination Product: REACH — The intervention consists of a mobility device called ActivLife developed by Alreh Medical, that is coupled with serious games, a Kinect sensor and a wearable sensor called Stepwatch, to continuously measure the patients physical activity.
  Arms: Intervention REACH group
Other: Standard of care — Standard of care for rehabilitation treatment for musculoskeletal patients.
  Arms: Control group (Standard of care)

SUMMARY:
Developed countries are facing the challenge of ageing societies, lack of infrastructure for healthcare and high cost of care. Researchers have been attempting to answer these problems by using innovative technology to promote healthy ageing. In this trial, the investigators test the efficiency and acceptance of a personal mobility device for elderly physical rehabilitation.

The main objective of the study is to investigate whether rehabilitation using the mobility equipment is as effective as the standard care; secondly, to determine if there is an improvement in clinical outcomes such as physical strength, balance, and risk of falls after using the mobility equipment; and third, to establish whether the use of the REACH concept adds value to the continuity of patient care, specifically in terms of engagement and motivation to be more active during the hospital stay and when returning home.

DETAILED DESCRIPTION:
The hospital-to-home transition is increasingly recognised as a critical period in the patient care, during which different incidents can occur and induce frequent re-hospitalisation. There is therefore a growing interest in strengthening the physical and functional capacities of hospitalised elderly patients to prevent re-hospitalisation.

Researchers have extensively studied the use of computer-aided physical rehabilitation to promote physical activity. Serious games coupled with monitoring devices such as Kinect have shown to positively impact patient's motivation to do rehabilitation exercises. Whether such devices would be as efficient as the standard care in the hospital and engage the elderly to remain active after discharge is still understudied.

In the present study , the researchers aim at conducting a randomised clinical trial with 46 patients during 6 weeks, to measure the added value of the REACH concept. REACH is a H2020 funded project, the project abbreviation stands for Responsive Engagement of the Elderly Promoting Activity and Customised Healthcare.

The intervention consists of a mobility device called ActivLife developed by Alreh Medical, that is coupled with serious games, a Kinect sensor and a wearable sensor called Stepwatch, to continuously measure the patients physical activity.

The main objective of the study is to investigate whether rehabilitation using the mobility equipment is as effective as the standard care; secondly, to determine if there is an improvement in clinical outcomes such as physical strength, balance, and risk of falls after using the mobility equipment; and third, to establish whether the use of the REACH concept adds value to the continuity of patient care, specifically in terms of engagement and motivation to be more active during the hospital stay and when returning home.

ELIGIBILITY:
Inclusion Criteria:

* seniors (65+) hospitalized in one of the involved sites at the Geneva University Hospital, with musculoskeletal issues (fracture, prosthesis, falls and low back pain), a minimal level of independence and strength (FIM >= 4 for the items regarding mobility and locomotion), and minimal level of cognitive ability (MMSE>=24); be able to interact with the equipment and be hospitalized at least 3 weeks at one of the hospitals.

Exclusion Criteria:

* patients that are considered too weak to interact with the device and that are hospitalized less than three weeks.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) Results | 6 weeks; (at the beginning of the intervention in the hospital and after 3 weeks when the participant is leaving the hospital, and after 3 additional weeks at home)
  Short Physical Performance Battery is a set of tests designed to measure functional status. and physical performance.
Change in Isometric Hand Grip Strength (IHGS) Results | 6 weeks; (at the beginning of the intervention in the hospital and after 3 weeks when the participant is leaving the hospital, and after 3 additional weeks at home)
  The purpose of the Isometric Hand Grip Strength test is to measure the maximum isometric strength of the hand and forearm muscles.

SECONDARY OUTCOMES:
Change in activity over 6 weeks | 6 weeks
  Measurement of activity level with stepwatch sensor. Continuous measurement of steps from participants with stepwatch sensor.

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Randriambelonoro M, Perrin Franck C, Herrmann F, Carmona GA, Geissbuhler A, Graf C, Frangos E. Gamified Physical Rehabilitation for Older Adults With Musculoskeletal Issues: Pilot Noninferiority Randomized Clinical Trial. JMIR Rehabil Assist Technol. 2023 Mar 6;10:e39543. doi: 10.2196/39543. PMID 36877563